CLINICAL TRIAL: NCT02161029
Title: Flexible Endoscopy Biopsies With the New Drill Biopsy Instrument for Submucous Tumors
Brief Title: Flexible Endoscopy Biopsies for Submucous Tumors With a New Drill Instrument
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Lund University Hospital (Other)
Responsible Party: Principal Investigator, Bruno Walther, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/97
Record Dates: First submitted 2014-03-25; First posted 2014-06-11 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Gastric Tumor
Keywords: Gastric tumor
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New drill biopsy instrument (Active Comparator): To take biopsies from gastric submucosal tumors with a new drill biopsy instrument used with flexible endoscopes.
  Interventions: Device: Flexible drill biopsy instrument
- Conventional biopsy instrument (Active Comparator): To take biopsies from gastric submucosal tumors with conventional biopsy forceps used with flexible endoscopes
  Interventions: Device: conventional biopsy instrument

INTERVENTIONS:
Device: Flexible drill biopsy instrument — Biopsies taken with the new drill biopsy instrument for flexible endoscopy
  Other Names: Endodrill (=Internal code name)
  Arms: New drill biopsy instrument
Device: conventional biopsy instrument — Biopsies taken with conventional biopsy forceps for flexible endoscopic instruments
  Arms: Conventional biopsy instrument

SUMMARY:
The purpose of this study is to determine whether the newly constructed CE (Conformité Européenne) marked drill biopsy instrument for flexible endoscopes can make possible representative biopsies of the increasing numbers of submucosal tumours in the gastrointestinal tract. The amount of submucous tissue ( micrograms and in % of all the biopsy) harvested with the new drill biopsy instrument used in flexible endoscopy investigations is measured in the study and compared to the amount of submucous tissue harvested with the existing biopsy forceps.

DETAILED DESCRIPTION:
Background: With the existing biopsy instruments for flexible endoscopy it's only possible to achieve superficial biopsies comprising the mucosa and very seldom some small fragments of the submucosa. It is, however, increasingly important to get biopsies from the submucous tissues because the tumors that are on the increase more than any other in the stomach is the GIST (GastroIntestinal Stroma Tumours) that grows in the submucosa. Cytology is not enough for a reliable diagnosis and to often not representative. Furthermore there is a well-known risk for tract seeding when sampling through the abdominal wall with a fine needle instrument.

The investigators have invented a new biopsy instrument for flexible endoscopy that is a drill within a cylinder that can be used for biopsies of the submucous tissues, for instance GIST-tumours, see www.BIBBInstruments.com.

Hypothesis: Will it be possible to achieve representative submucous tissue from the gastrointestinal tract with the newly constructed drill biopsy instrument for flexible endoscopy. The investigators hypothesize that the amount of tissue harvested with the new drill biopsy instrument will give significantly more amount of tissue to evaluate for the pathologist than the existing biopsy forceps.

Method: Ten patients with tumours in the submucosa of the stomach are examined with a gastroscope. The investigator decides where the first biopsy should be taken and randomly the investigator blindly get the new drill instrument or the conventional biopsy forceps and take the biopsy on the decided localization. The next site of the tumour is decided and again blindly the investigator get one of the two biopsy instruments according to a previously decided scheme. Six biopsies (three with each of the two biopsy tools) in every patient are harvested in ten patients. With altogether 30 specimen for each biopsy instrument and a difference of 1/3 which is a low calculated difference 10 patients as above will give a 80 % Power (Chi-2 = 5.40, p = 0.02*). The amount of submucous tissue harvested with the two biopsy instruments are measured in microgram and as percentage of all the biopsy and compared. The quality of the specimens are also calculated.

ELIGIBILITY:
Inclusion Criteria:

* Submucous gastrointestinal tumours

Exclusion Criteria:

* No gastrointestinal submucous tumor
* Submucosal hemangioma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2015-03-27 (Actual); Study Completion 2015-03-27 (Actual)

PRIMARY OUTCOMES:
Amount of submucous tissue in gastrointestinal submucosal tumors harvested with a new drill biopsy instrument used with flexible endoscopes. | Within 30 days for each patient
  Amount of submucous tissue adequate for histological examination harvested with the new drill biopsy instrument for flexible endoscopy and compared to the amount harvested with the existing biopsy forceps in a randomized setting.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno S Walther, MD, Principal Investigator — Professor
Locations (1):
- Department of Surgery, Lund University, Lund, Sweden

REFERENCES:
- See also: Related Info — http://www.Bibbinstruments.com